CLINICAL TRIAL: NCT06080451
Title: Implementing Integrated Diabetes and Hypertension Management in Guatemala Using the HEARTS Model
Brief Title: Implementing HEARTS in Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Institute of Nutrition of Central America and Panama (Other); Ministry of Health, Guatemala (Other Government)
Responsible Party: Principal Investigator, David Flood, Assistant Professor of Medicine, University of Michigan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00234613; K23HL161271 (NIH)
Record Dates: First submitted 2023-10-06; First posted 2023-10-12 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Cardiovascular Diseases | interventions — Heart, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEARTS implementation - Patients (Experimental): A trial for 6 months will be carried out in 11 Ministry of Health primary care facilities starting in October 2023. This arm consists of the patients whose health markers will be monitored through the study.
  Interventions: Other: Integrated Diabetes and Hypertension Primary Care Model
- HEARTS implementation - Providers (Experimental): A trial for 6 months will be carried out in 11 Ministry of Health primary care facilities starting in October 2023. This arm consists of the health care providers who will be administering care to the patient participants.
  Interventions: Other: Integrated Diabetes and Hypertension Primary Care Model - Providers

INTERVENTIONS:
Other: Integrated Diabetes and Hypertension Primary Care Model — The intervention consists of five components that align with the World Health Organization Technical Package for Cardiovascular Disease Management in primary Health Care.
  1. Training health workers on diabetes and hypertension treatment protocols
  2. Team-based care and task sharing
  3. Strengthening access to medications and diagnostics
  4. Electronic medical record system and registry
  5. Systems monitoring and feedback of key indicators
  Other Names: HEARTS
  Arms: HEARTS implementation - Patients
Other: Integrated Diabetes and Hypertension Primary Care Model - Providers — The intervention consists of five components that align with the World Health Organization Technical Package for Cardiovascular Disease Management in primary Health Care.
  1. Training health workers on diabetes and hypertension treatment protocols
  2. Team-based care and task sharing
  3. Strengthening access to medications and diagnostics
  4. Electronic medical record system and registry
  5. Systems monitoring and feedback of key indicators
  Health care providers will administer this intervention to patient participants and will report on their experience.
  Arms: HEARTS implementation - Providers

SUMMARY:
The HEARTS Technical Package was developed by the World Health Organization to address the implementation gap of cardiovascular disease prevention in low- and middle-income countries. Guatemala is a middle-income country that is currently implementing HEARTS. National authorities are interested in exploring how hypertension and diabetes management can be integrated in HEARTS implementation. The objective of this study is to conduct a feasibility and acceptability pilot trial of integrated hypertension and diabetes management based on HEARTS in the publicly funded primary care system in Guatemala.

DETAILED DESCRIPTION:
A single-arm pilot trial for 6 months will be carried out in 11 Ministry of Health primary care facilities starting in September 2023. A planned sample of 100 adult patients diagnosed with diabetes (n=45), hypertension (n=45), or both (n=10) will be enrolled. The intervention will consist of HEARTS-aligned components: Training health workers on Healthy-lifestyle counseling and Evidence-based treatment protocols; strengthening Access to medications and diagnostics; training on Risk-based cardiovascular disease management; Team-based care and task sharing; and Systems monitoring and feedback, including implementation of a facility-based electronic monitoring tool at the individual level. Co-primary outcomes of feasibility and acceptability will be assessed using an explanatory sequential mixed methods design. Secondary outcomes include clinical effectiveness (treatment with medication, glycemic control, and blood pressure control) and key implementation outcomes (adoption, fidelity, usability, and sustainability).

ELIGIBILITY:
Patient participants

Inclusion criteria:

* Non-pregnant adults aged ≥18 years
* Diagnoses of type 2 diabetes or hypertension
* Present for routine care at participating MOH primary health facilities

Exclusion criteria:

* Confirmed or suspected type 1 diabetes
* Pregnant
* Are not managed at MOH health centers or health posts

Provider/other participants

Inclusion criteria:

• Participation in delivering HEARTS or on the Technical Advisory Committee

Exclusion criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Flood, MD, Principal Investigator — University of Michigan
Locations (1):
- Ministry of Health clinics, San Pablo La Laguna, Departamento de Sololá, Guatemala

IPD SHARING:
Plan to Share IPD: Yes
This project will produce multiple types of data, including patients' clinical information, health facility assessments, and structured and semi-structured interviews. Deidentified data, analytic code, and data dictionaries will be made available on the NHLBI Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) data repository (https://biolincc.nhlbi.nih.gov/) after the study concludes. Semi-structured interview transcripts and structured questionnaire data will not be shared due to privacy concerns and risk for re-identification.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Wellmann IA, Ayala LF, Rodriguez JJ, Guetterman TC, Irazola V, Palacios E, Huffman MD, Rohloff P, Heisler M, Ramirez-Zea M, Flood D. Implementing integrated hypertension and diabetes management using the World Health Organization's HEARTS model: protocol for a pilot study in the Guatemalan national primary care system. Implement Sci Commun. 2024 Jan 9;5(1):7. doi: 10.1186/s43058-023-00539-8. PMID 38195600
- [Result] Wellmann IA, Ayala LF, Valley TM, Irazola V, Huffman MD, Heisler M, Rohloff P, Donis R, Palacios E, Ramirez-Zea M, Flood D. Evaluating the World Health Organization's Hearts Model for Hypertension and Diabetes Management: A Pilot Implementation Study in Guatemala. Glob Heart. 2025 Jan 31;20(1):9. doi: 10.5334/gh.1397. eCollection 2025. PMID 39896314

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Providers not considered Enrolled
Period: Overall Study
Arm/Group | HEARTS Implementation - Patients | HEARTS Implementation - Providers
Started | 964 | 40 (Providers trained on the intervention)
Completed Provider Survey (Not Applicable to Patient Arm) | 0 | 20
Completed | 964 | 20
Not Completed | 0 | 20

BASELINE CHARACTERISTICS:
Groups:
- HEARTS Implementation - Patients: A trial for 6 months will be carried out in 11 Ministry of Health primary care facilities starting in October 2023. This arm consists of the patients whose health markers will be monitored through the study.
  Integrated Diabetes and Hypertension Primary Care Model: The intervention consists of five components that align with the World Health Organization Technical Package for Cardiovascular Disease Management in primary Health Care.
  1. Training health workers on diabetes and hypertension treatment protocols
  2. Team-based care and task sharing
  3. Strengthening access to medications and diagnostics
  4. Electronic medical record system and registry
  5. Systems monitoring and feedback of key indicators
- HEARTS Implementation - Providers: A trial for 6 months will be carried out in 11 Ministry of Health primary care facilities starting in October 2023. This arm consists of the health care providers who will be administering care to the patient participants.
  Integrated Diabetes and Hypertension Primary Care Model - Providers: The intervention consists of five components that align with the World Health Organization Technical Package for Cardiovascular Disease Management in primary Health Care.
  1. Training health workers on diabetes and hypertension treatment protocols
  2. Team-based care and task sharing
  3. Strengthening access to medications and diagnostics
  4. Electronic medical record system and registry
  5. Systems monitoring and feedback of key indicators
  Health care providers will administer this intervention to patient participants and will report on their experience.
- Total: Total of all reporting groups
Arm/Group | HEARTS Implementation - Patients | HEARTS Implementation - Providers | Total
Number analyzed (Participants) | 964 | 20 | 984
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Age data was only collected for the patient arm and not for the provider arm.
  years
    number analyzed (Participants) | 964 | 0 | 964
    (all) | 55.2 [44.1 to 66.1] |  | 55.2 [44.1 to 66.1]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data was only collected for the patient arm and not for the provider arm.
  Participants
    number analyzed (Participants) | 964 | 0 | 964
    Female | 760 |  | 760
    Male | 204 |  | 204
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data was only collected for the patient arm and not for the provider arm.
  Participants
    number analyzed (Participants) | 964 | 0 | 964
    Hispanic or Latino | 474 |  | 474
    Not Hispanic or Latino | 486 |  | 486
    Unknown or Not Reported | 4 |  | 4
Region of Enrollment [Number; unit: participants]
  Guatemala | 964 | 20 | 984

OUTCOME MEASURES:

1. Primary Outcome: Score on Feasibility of Intervention Measure (FIM) Questionnaire
Description: Feasibility will be assessed among Ministry of Health (MOH) participants through the four-item Feasibility of Intervention Measure (FIM) Questionnaire and semi-structured interviews. A Spanish-language version of the FIM will be adapted for this project. Scores will be on a scale of 1 to 5, with 1 being the worst and 5 being the best. The average score for each participant will be used.
Time Frame: 6 months
Population: This outcome measure only applies to the Providers group. No data was collected for the Patients group. Only 20 providers responded to this survey.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HEARTS Implementation - Providers
Number analyzed (Participants) | 20
score on a scale | 5.0 [5.0 to 5.0]

2. Primary Outcome: Number of Target Health Districts That Met Enrollment Goals
Description: This study will be working with two different health districts, one in the west and the other in the east. This measure is the number of districts that met enrollment goals for patients for patients with diabetes (at least 25) and also for patients with hypertension (at least 25). A given patient may have both diabetes and hypertension and thus count toward each benchmark
Time Frame: 6 months
Population: This outcome measure only applies to the Patients group. No data was collected for the Providers group.
Measure: Count of Units; unit: Districts
Units Other Than Participants: Districts
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 964
Number analyzed (Districts) | 2
Districts | 2

3. Primary Outcome: Score on Acceptability of Intervention Measure (AIM) Questionnaire
Description: Acceptability will be assessed among providers through the four-item Acceptability Intervention Measure (AIM) Questionnaire and semi-structured interviews. A Spanish-language version of the AIM will be adapted for this project. Scores will be on a scale of 1 to 5, with 1 being the worst and 5 being the best. The average score for each participant will be used.
Time Frame: 6 months
Population: Only 20 providers responded to this survey. This measure only applies to the provider arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HEARTS Implementation - Providers
Number analyzed (Participants) | 20
score on a scale | 5.0 [4.8 to 5.0]

4. Primary Outcome: Proportion of Patient Participants With Subsequent Follow-up Visit Within 3 Months
Description: Proportion of patient participants with subsequent follow-up visit within 3 months in both regions combined.
Time Frame: 3 months
Measure: Number; unit: percentage of patients
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 964
percentage of patients | 36

5. Secondary Outcome: Hypertension Treatment Rate
Description: Number of patients receiving hypertension medication treatment in the 6th month of the study.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 964
Participants | 197

6. Secondary Outcome: Diabetes Treatment Rate
Description: Number of patients receiving diabetes medication treatment in the 6th month of the trial..
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 964
Participants | 108

7. Secondary Outcome: Proportion of Patient Participants Achieving Glycemic Control
Description: Proportion achieving glycemic control (fasting blood glucose <115 mg/dl or random blood glucose <160 mg/dl) among patients with diabetes
Time Frame: 6 months
Population: Monitoring system only captured data from 39 participants and failed to capture data for other participants
Measure: Number; unit: percent
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 39
percent | 41

8. Secondary Outcome: Proportion Achieving Control of Blood Pressure
Description: Proportion achieving control of blood pressure (<130/80 mmHg) among patients with hypertension. This information will be taken from electronic medical records.
Time Frame: 6 months
Population: The monitoring system was incompletely utilized and only captured this data for 83 participants
Measure: Number; unit: percent
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 83
percent | 50.6

9. Secondary Outcome: Adoption
Description: Count and percentage of participating health facilities who enrolled at least one patient with hypertension or diabetes.
Time Frame: 6 months
Population: One of the eleven initially planned health facilities declined to participate in the study.
Measure: Count of Units; unit: Clinics
Units Other Than Participants: Clinics
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 964
Number analyzed (Clinics) | 10
Clinics | 10

10. Secondary Outcome: Fidelity - Health Worker Training
Description: Number of health workers in each district attending all training sessions
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | HEARTS Implementation - Providers
Number analyzed (Participants) | 40
Participants
  District 1 | 20
  District 2 | 20

11. Secondary Outcome: Fidelity - Team-based Care and Task Sharing
Description: Proportion of primary health facilities conducting at least one care coordination meeting
Time Frame: 6 months
Population: This group is of Clinics, not of participants. One of the eleven initially planned facilities declined to participate in this study.
Measure: Count of Units; unit: Clinics
Units Other Than Participants: Clinics
Groups:
- HEARTS Implementation - Clinics: A trial for 6 months will be carried out in 11 Ministry of Health primary care facilities starting in October 2023. This group consists of the clinics at which the patient participants will be receiving care from the provider participants.
Arm/Group | HEARTS Implementation - Clinics
Number analyzed (Participants) | NA
Number analyzed (Clinics) | 10
Clinics | 10

12. Secondary Outcome: Fidelity - Access to Medicines and Diagnostics
Description: Months in which primary health facilities had monthly availability of Ministry of Health medications and diagnostics for diabetes and hypertension. Drugs include antihypertensive medications (hydrochlorothiazide, enalapril, losartan) and oral hypoglycemic agents (metformin and glimepiride). Diagnostics including blood pressure cuffs and monitors, glucometers, lancets, and glucose strips.
  Data is reported in "clinic-months", which is the sum number of months that each clinic reported monthly availability of medications and diagnostics (n=60 total clinic months(10 clinics x 6 months)).
Time Frame: 6 months
Population: One of the eleven initially planned facilities declined to participate in this study.
Measure: Number; unit: clinic-months
Units Other Than Participants: Clinics
Groups:
- HEARTS Implementation - Clinics: A trial for 6 months will be carried out in 11 Ministry of Health primary care facilities starting in October 2023. This arm consists of the clinics at which the patient participants received care from the provider participants.
Arm/Group | HEARTS Implementation - Clinics
Number analyzed (Participants) | NA
Number analyzed (Clinics) | 10
clinic-months | 49

13. Secondary Outcome: Fidelity - Facility-based Electronic Monitoring Tool
Description: Proportion of patient visits captured in DHIS2 during the study compared to comprehensive records in the Ministry of Health's Health Management Information System. Data was collected at the end of the 6th month study. Data is presented as percent of visits that were captured.
Time Frame: 6 months
Population: Number of patient visits
Measure: Number; unit: percentage of visits
Units Other Than Participants: Visits
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 964
Number analyzed (Visits) | 1374
percentage of visits | 7.6

14. Secondary Outcome: Usability
Description: Average score on the System Usability Scale questionnaire. Scores have a range of 0 (worst) to 100 (best). Questionnaire was given to the provider arm only.
Time Frame: 6 months
Population: Questionnaire was given to the provider arm only. 20 of the 40 providers responded to this survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HEARTS Implementation - Providers
Number analyzed (Participants) | 20
units on a scale | 67.7 (23.5)

15. Secondary Outcome: Sustainability
Description: Mean score on a sustainability questionnaire. Questionnaire was created by combining 6 questions from the Program Sustainability Assessment Tool (PSAT) and Clinical Sustainability Assessment Tools (CSAT). Scores range from 1 (worst) to 7 (best). The data reported is the median of the mean scores for each of the health providers.
Time Frame: 6 months
Population: 20 of the 40 provider participants responded to this survey.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | HEARTS Implementation - Providers
Number analyzed (Participants) | 20
units on a scale | 5.3 [4.8 to 5.9]

16. Secondary Outcome: Mean Systolic Blood Pressure
Description: Mean systolic blood pressure among patients with hypertension
Time Frame: 6 months
Population: While this outcome measure was part of the original plan for the study, implementation of monitoring this outcome failed and data was only collected for 72 patients. This outcome measure did not apply to the provider's arm.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 72
mmHg | 141.7 (18.5)

17. Secondary Outcome: Mean Diastolic Blood Pressure
Description: Mean diastolic blood pressure among patients with hypertension
Time Frame: 6 Months
Population: While this outcome measure was part of the original plan for the study, implementation of monitoring this outcome failed and data was only collected for 71 patients. This outcome measure did not apply to the provider's arm. While Systolic pressure was recorded for 72 participants, diastolic pressure was not recorded from one of these participants due to an unknown error at the clinic.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 71
mmHg | 81.5 (11.2)

18. Secondary Outcome: Fidelity - Chart Audit
Description: Proportion of clinical visits that are guideline concordant according to study team's audit of least 25% of patient visits
Time Frame: 6 months
Population: While this outcome measure was part of the original plan for the study, implementation of monitoring this outcome failed and no data was collected due to physicians' declination to use the software. This measure only applied to the patients arm.
Arm/Group | HEARTS Implementation - Patients
Number analyzed (Participants) | 0

19. Secondary Outcome: Fidelity - Systems Monitoring and Feedback
Description: Proportion of quarterly reports viewed by health district administrators
Time Frame: 6 months
Population: While this outcome measure was part of the original plan for the study, implementation of monitoring this outcome failed and no data was collected due to physicians' declination to use the software.
Arm/Group | HEARTS Implementation - Patients | HEARTS Implementation - Providers
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Providers were asked to provide patient adverse event information to the Michigan team when they occurred. No reports were sent.
  No adverse event data collection was planned for the provider arm.
Arm/Group | HEARTS Implementation - Patients | HEARTS Implementation - Providers
All-Cause Mortality (participants affected / at risk) | 0/964 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/964 | 0/0
Other Adverse Events (participants affected / at risk) | 0/964 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/51/NCT06080451/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT06080451/ICF_001.pdf